CLINICAL TRIAL: NCT07063043
Title: Clinical Research on 68Ga-FAPI PET/CMR in Cardiovascular Diseases
Status: Recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025YS-039
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases (CVD)
Keywords: Cardiovascular diseases; FAPI; PET/MR
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Research group: Thirty patients with cardiovascular diseases were enrolled as the research group.
- Healthy controls: Ten healthy individuals were enrolled as the healthy controls.

SUMMARY:
FAP-targeted PET imaging using 68Ga-FAPI enables early detection of myocardial fibrosis. Combined PET/CMR provides comprehensive cardiac assessment without extra radiation. This advanced imaging approach improves diagnosis and personalized treatment for better patient outcomes.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) are among the leading causes of death and disability worldwide. According to statistics from the World Health Organization (WHO), over 17 million people die from CVDs each year, accounting for 31% of global mortality[1]. In China, the incidence and mortality rates of CVDs continue to rise alarmingly. The China Cardiovascular Health and Diseases Report indicates that approximately 300 million Chinese suffer from CVDs, with annual CVD-related deaths exceeding 4 million - representing over 40% of the country's total deaths[2]. These concerning trends highlight CVDs as a major public health crisis demanding urgent attention.

Recent advances in molecular imaging have opened new avenues for CVD diagnosis and management. Fibroblast activation protein (FAP), a type II transmembrane serine protease, shows minimal expression in normal tissues but becomes markedly upregulated in various pathological conditions including malignant tumors, inflammatory diseases, and fibrotic processes[3,4]. Of particular significance is its role in myocardial fibrosis - a key pathological mechanism underlying many CVDs[5]. Current diagnostic methods for myocardial fibrosis remain limited, with histopathology being invasive and conventional imaging techniques like echocardiography and cardiac MR (CMR) only detecting late-stage changes. The emergence of radiolabeled FAP inhibitors (FAPIs) has enabled non-invasive visualization of early myocardial fibrosis, offering unprecedented opportunities for dynamic monitoring of disease progression and treatment response.

The clinical potential of FAPI-based imaging in CVDs is increasingly recognized. Although still in the exploratory phase, studies have consistently demonstrated FAPI uptake in various CVD animal models and human patients, confirming the activation of cardiac fibroblasts and FAP expression across different disease states. This technology provides three key advantages: first, it allows in vivo visualization of fibroblast activity at molecular levels; second, it enables early detection of fibrotic changes before structural damage occurs; third, when combined with other imaging modalities, it permits comprehensive assessment of disease progression. These capabilities make FAPI imaging a powerful tool for identifying candidates for anti-fibrotic therapy and monitoring treatment efficacy.

Integrated PET/MR technology represents another major breakthrough in cardiac imaging. By combining the superior soft-tissue resolution of MR with PET's molecular sensitivity, simultaneous PET/CMR systems provide unparalleled insights into cardiac structure and function[6]. This hybrid approach integrates anatomical details from CMR (including late gadolinium enhancement patterns) with metabolic information from PET, delivering more comprehensive data than either modality alone. Importantly, PET/CMR achieves this without additional radiation exposure from CT components, making it particularly suitable for longitudinal studies. While clinical applications in CVDs remain investigational, PET/CMR holds tremendous promise for advancing our understanding of disease mechanisms and enabling personalized treatment strategies.

This research project aims to harness these technological advancements for improved CVD management. By implementing 68Ga-FAPI PET/CMR multi-modal imaging, we seek to achieve precise quantification of myocardial fibrosis and comprehensive evaluation of cardiac function in a single examination. The synergistic combination of 68Ga-FAPI's molecular targeting capability with CMR's structural and functional assessment offers several clinical benefits: it streamlines diagnostic workflows, enhances accuracy, facilitates timely intervention, and ultimately may improve patient outcomes. Through this innovative approach, we hope to establish a new paradigm in CVD care that combines cutting-edge imaging technology with personalized medicine principles, thereby addressing the growing burden of cardiovascular diseases more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed clinical diagnosis of cardiovascular disease by a cardiologist, based on genetic testing, family history, and comprehensive clinical evaluation including physical examination, echocardiography, and when indicated, cardiac MRI findings.
* Age requirement: >18 years.
* Patients should demonstrate stable cardiovascular status without significant changes in symptoms, treatment, or clinical findings for a specified pre-enrollment period.
* Participants must be capable of providing informed consent and willing to adhere to all study requirements, including follow-up procedures.

Exclusion Criteria:

* History of malignancy
* Documented cardiovascular diseases, including coronary artery disease, myocardial infarction, or related conditions
* Implanted metallic devices (e.g., pacemakers, aneurysm clips) or other MRI-incompatible medical prostheses
* Claustrophobia
* Pregnancy or lactation
* Known hypersensitivity to gadolinium-based contrast agents
* Renal impairment (eGFR <30 mL/min/1.73m² by CKD-EPI equation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cardiovascular diseases
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
CE-CMR | After the patient completes the scan, an average of 2 days.
  Left ventricular wall thickness was quantified on short-axis cine images using the MR cardiac analysis software .
CE-MRI | After the patient completes the scan, an average of 2 days.
  Left ventricular ejection fraction (LVEF) was calculated from short-axis cine images using the cardiac MR analysis software.
PET | After the patient completes the scan, an average of 2 days.
  The maximum standardized uptake value (SUVmax) was calculated for each myocardial segment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
For the protection of patient privacy, we will not share patient information, but other researchers can apply through the project contact person if they have reasonable reasons.